CLINICAL TRIAL: NCT05169996
Title: Development and Evaluation of a Virtual Reality Puzzle Game to Decrease Food Intake
Brief Title: Virtual Reality Effects on Food Intake Game to Decrease Food Intake
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tilburg University (Other)
Responsible Party: Principal Investigator, Laura Nynke van der Laan, Associate professor, Tilburg University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2018-PC-9033
Record Dates: First submitted 2021-11-26; First posted 2021-12-27 (Actual); Last update posted 2021-12-27 (Actual); Status verified 2021-12

CONDITIONS: Food Intake
Keywords: virtual reality; pre-exposure; food cravings

STUDY DESIGN:
Intervention Model Description: In a 2 (game: real vs virtual) x 2 (product: food vs non-food) between-subjects design lab experiment, the effectiveness of pre-exposure to food in a VR game is tested. A fifth condition was added ("VR x branded food") in order to examine brand effects.
Who Masked: Participant
Masking Description: Participants were not informed about in which arm of the study they were allocated.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Real Food (Experimental): Participants are exposed to a tangram game with puzzle pieces from chocolate.
  Interventions: Other: Real Food
- Real Nonfood (Experimental): Participants are exposed to a tangram game with puzzle pieces from wood.
  Interventions: Other: Real Nonfood
- Virtual reality Food (Experimental): Participants are exposed to a virtual reality experience with a tangram game with puzzle pieces from (virtual) chocolate.
  Interventions: Other: Virtual reality Food
- Virtual reality Nonfood (Experimental): Participants are exposed to a virtual reality experience with a tangram game with puzzle pieces from (virtual) wood.
  Interventions: Other: Virtual reality Nonfood
- Virtual reality Food Branded (Experimental): Participants are exposed to a virtual reality experience with a tangram game with puzzle pieces from (virtual) chocolate. In the background of the puzzle, a brand is shown.
  Interventions: Other: Virtual reality Food Branded

INTERVENTIONS:
Other: Real Food — The game was played while sitting behind a table in the lab. The task in the game was to finish a tangram puzzle. In the Real Food condition, the tangram pieces were tempting food products (i.e., pieces of chocolate). Players had to physically move the chocolate pieces with their hands and puzzle them together.
  Arms: Real Food
Other: Real Nonfood — The game was played while sitting behind a table in the lab. The task in the game was to finish a tangram puzzle. In the Real Nonfood condition, the tangram pieces were plain pieces (i.e., pieces of wood). Players had to physically move the wooden pieces with their hands and puzzle them together.
  Arms: Real Nonfood
Other: Virtual reality Food — The game was played by wearing a VR head-mounted display (HMD VR: HTC Vive) and people could interact in the virtual environment with the hand-held controllers. The task in the game was to finish a tangram puzzle. In the Virtual Reality Food condition, the tangram pieces were tempting food products (i.e., pieces of virtual chocolate). Players had to physically move the virtual chocolate pieces with the grab button on the controller and puzzle them together.
  Arms: Virtual reality Food
Other: Virtual reality Nonfood — The game was played by wearing a VR head-mounted display (HMD VR: HTC Vive) and people could interact in the virtual environment with the hand-held controllers. The task in the game was to finish a tangram puzzle. In the Virtual Reality Nonfood condition, the tangram pieces were plain pieces (i.e., pieces of virtual wood). Players had to physically move the virtual wood pieces with the grab button on the controller and puzzle them together.
  Arms: Virtual reality Nonfood
Other: Virtual reality Food Branded — The game was played by wearing a VR head-mounted display (HMD VR: HTC Vive) and people could interact in the virtual environment with the hand-held controllers. The task in the game was to finish a tangram puzzle. In the Virtual Reality Food condition, the tangram pieces were tempting food products (i.e., pieces of virtual chocolate). Players had to physically move the virtual chocolate pieces with the grab button on the controller and puzzle them together. In the background of the puzzle, a chocolate brand ('Milka') is shown
  Arms: Virtual reality Food Branded

SUMMARY:
Aims:

* The first aim was to replicate the pre-exposure effect. This was done by assessing the effect of exposing participants to a puzzle game with real foods compared to real nonfoods on food intake.
* The second aim was to investigate the potential of VR for eliciting the pre-exposure effect. This was done by comparing the effect of a VR puzzle game with foods to a VR puzzle game with nonfoods on food intake.
* The third aim was to assess the effect of branding in VR on brand responses and the role of emotional responses herein. This was done by comparing a branded virtual puzzle game with foods with a (non-branded) virtual puzzle game with foods.

Study design: a randomized 2 (game: real vs virtual) x 2 (product: food vs non-food) between-subjects design lab experiment, the effectiveness of pre-exposure to food in a VR game is tested. A fifth condition was added ("VR x branded food") in order to examine brand effects.

DETAILED DESCRIPTION:
Aim: Every day, people are exposed to a wide variety of tasty foods, which is thought to be the leading cause of overeating. However, subsequent intake is believed to decrease when individuals engage with foods outside an eating context in an unrelated task-this is called the pre-exposure effect. Thus far, this effect has only been found when tempting foods are physically present. The current study aims to examine whether the effect also occurs when hyper-realistic food is present in VR.

Virtual reality (VR) provides the ultimate level of immersion, creating a sense of physical presence in the three-dimensional virtual environment. Therefore, VR has a major potential for implementation of the pre-exposure effect in an intervention and to assess the underlying psychological mechanisms. The level of immersion is also thought to increase the effects of brand exposure. Here, a VR game was developed with realistic virtual foods and it was assessed in the lab whether interaction with virtual foods decreases subsequent food intake similarly as real foods do. In addition the effects of brand exposure in VR on brand-relevant outcomes were assessed.

Aims:

* The first aim was to replicate the pre-exposure effect. This was done by assessing the effect of exposing participants to a puzzle game with real foods compared to real nonfoods on food intake.
* The second aim was to investigate the potential of VR for eliciting the pre-exposure effect. This was done by comparing the effect of a VR puzzle game with foods to a VR puzzle game with nonfoods on food intake.
* The third aim was to assess the effect of branding in VR on brand responses and the role of emotional responses herein. This was done by comparing a branded virtual puzzle game with foods with a (non-branded) virtual puzzle game with foods.

Study design: In a randomized 2 (game: real vs virtual) x 2 (product: food vs non-food) between-subjects design lab experiment, the effectiveness of pre-exposure to food in a VR game is tested. A fifth condition was added ("VR x branded food") in order to examine brand effects.

ELIGIBILITY:
Inclusion Criteria:

* None (except for age 18-30)

Exclusion Criteria:

* Peanut allergy (self-reported)

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 202 (Actual)
Dates: Start 2018-05-09 (Actual); Primary Completion 2018-09-26 (Actual); Study Completion 2018-09-26 (Actual)

PRIMARY OUTCOMES:
Food intake | During the lab session
  Food intake (chocolates) in grams was measured by weighting the bowls of the taste test
Brand attitude | During the lab session
  Brand attitude was measured using a six-item 7-point semantic differential scale ranging from 1 (i.e., 'bad', 'unappealing', 'unpleasant', 'unattractive', 'boring', 'dislike') to 7 ('good', 'appealing', 'pleasant', 'attractive', 'exciting', 'like'), with the item "Select the answers that best reflect your opinion of the chocolate brand Milka"
Purchase intention | During the lab session
  Purchase intention was measured on a single-item 7-point scale ranging from 1 ('totally disagree') to 7 ('totally agree') by asking the participants to indicate how much they agreed with the statement "I am planning on buying Milka chocolate within the next seven days."

SECONDARY OUTCOMES:
Virtual product appeal | During the lab session
  One question was asked to measure virtual product appeal: 'How appealing was the chocolate you saw while playing the game?' This questions was answered on a visual analog scale ranging from 0 ('not appealing at all') to 100 ('extremely appealing').
Craving for virtual chocolate | During the lab session
  One question was asked to measure craving for virtual chocolate: 'How much did you feel like eating the chocolate?'. This questions was answered on a 7-point scale ranging from 1 ('Not at all') to 7 ('A whole lot')
Emotional response | During the lab session
  The self-assessment manikin (SAM) scales (Bradley & Lang, 1994) were used for measuring emotional responses. For this self-reported measure of emotional response, participants were shown a row of five manikins per emotional dimension that differed in the level of arousal or valence they portrayed. For the scale measuring arousal, the first manikin seemed very calm, but the final one seemed very excited. Similarly, for the scale measuring valence, the first manikin seemed very sad, and the final one seemed very happy. The participants were asked to indicate their emotional state while playing the VR game on a 9-point response scale. Each odd number of the scale corresponded with one of the five manikins for arousal and valence.
Perceived entertainment value | During the lab session
  Perceived entertaining value of the game was measured using a four-item 7-point scale ranging from 1 ('totally disagree') to 7 ('totally agree') (Martí-Parreno, Aldas-Manzano, Curras-Perez, & Sanchez-García, 2013) with the following items: 'Playing the game has been enjoyable', 'I had fun playing the game', 'Playing the game has been pleasurable ', and 'Playing the game has been exciting '.
Game difficulty | During the lab session
  Game difficulty was measured using a four-item ('To what extent did you find the game easy', 'To what extent did you feel like you were making progress towards the end of the game?', 'How well do you think you performed in the game?', and 'To what extent did you find the game challenging?') 7-point scale ranging from 1 ('not at all') to 7 ('very much so').

CONTACTS AND LOCATIONS:
Overall Officials: Laura Nynke Laura Nynke, Dr. Ir., Principal Investigator — Tilburg University
Locations (1):
- University of Amsterdam - ComLab, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Liu Y, Stamos A, Dewitte S, van Berlo ZMC, van der Laan LN. Development and Evaluation of a Virtual Reality Puzzle Game to Decrease Food Intake: Randomized Controlled Trial. JMIR Serious Games. 2022 Feb 3;10(1):e31747. doi: 10.2196/31747. PMID 35113028